CLINICAL TRIAL: NCT00036738
Title: Allogeneic Nonmyeloablative Hematopoietic Stem Cell Transplant for Patients With BCR-ABL Tyrosine Kinase Inhibitor Responsive Ph+ Acute Leukemia ? A Multi-center Trial
Brief Title: Fludarabine Phosphate and Total-Body Irradiation Followed by Donor Peripheral Blood Stem Cell Transplant in Treating Patients With Acute Lymphoblastic Leukemia or Chronic Myelogenous Leukemia That Has Responded to Treatment With Imatinib Mesylate, Dasatinib, or Nilotinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1581.00; NCI-2010-00131 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1581.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA078902 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Results first posted 2017-08-22 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2019-12

CONDITIONS: Adult Acute Lymphoblastic Leukemia in Remission; Adult B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1; Blastic Phase; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Phase of Disease; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Disease
MeSH Terms: conditions — Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — Cyclosporine; Cyclosporins; Dasatinib; fludarabine phosphate; Imatinib Mesylate; Mycophenolic Acid; nilotinib; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (allogeneic nonmyeloablative HSCT) (Experimental): See Detailed Description
  Interventions: Drug: Cyclosporine; Drug: Dasatinib; Drug: Fludarabine Phosphate; Drug: Imatinib Mesylate; Drug: Mycophenolate Mofetil; Drug: Nilotinib; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation; Biological: Therapeutic Allogeneic Lymphocytes; Radiation: Total-Body Irradiation

INTERVENTIONS:
Drug: Cyclosporine — Given IV or PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Sprycel
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Drug: Imatinib Mesylate — Given PO
  Other Names: CGP 57148; CGP57148B; Gleevec; Glivec; STI 571; STI-571; STI571
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Drug: Nilotinib — Given PO
  Other Names: AMN 107; Tasigna
Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation — Undergo nonmyeloablative allogeneic PBSC transplantation
  Other Names: Non-myeloablative allogeneic transplant; Nonmyeloablative Stem Cell Transplantation; NST
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic PBSC transplantation
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Biological: Therapeutic Allogeneic Lymphocytes — Given IV
  Other Names: Allogeneic Lymphocytes
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: Total Body Irradiation; Whole-Body Irradiation

SUMMARY:
This phase II trial is studying how well fludarabine phosphate and total-body irradiation followed by donor peripheral blood stem cell transplant work in treating patients with acute lymphoblastic leukemia or chronic myelogenous leukemia that has responded to previous treatment with imatinib mesylate, dasatinib, or nilotinib. Giving low doses of chemotherapy, such as fludarabine phosphate, and total-body irradiation (TBI) before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Giving an infusion of the donor's T cells (donor lymphocyte infusion) after the transplant may help increase this effect. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving mycophenolate mofetil and cyclosporine after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the rate of leukemia relapse can be decreased for patients with chronic myelogenous leukemia in blast crisis (CML-BC) and Philadelphia chromosome positive acute lymphoblastic leukemia (Ph+ ALL) responsive to imatinib mesylate (or either dasatinib or nilotinib for patients who have imatinib-resistant disease or who are intolerant of imatinib) followed by nonmyeloablative hematopoietic stem cell transplantation (HSCT) compared to historical controls given high-dose conventional allogeneic HSCT or chemotherapy.

II. To determine whether the rate of transplantation-related mortality (TRM) can be decreased for patients with CML-BC and Ph+ ALL responsive to imatinib mesylate (or dasatinib or nilotinib) followed by nonmyeloablative HSCT compared to historical controls given high-dose conventional allogeneic HSCT or chemotherapy.

SECONDARY OBJECTIVES:

I. To evaluate whether donor lymphocyte infusion (DLI) can be safely used in patients with mixed or full donor chimerism as preemptive therapy to eliminate minimal residual disease.

OUTLINE:

INDUCTION THERAPY: Patients continue to receive imatinib mesylate orally (PO), dasatinib PO, or nilotinib PO once or twice daily until day -2 and resume on day 14 or when blood counts recover after peripheral blood stem cell (PBSC) transplantation.

NONMYELOABLATIVE CONDITIONING: Patients receive fludarabine intravenously (IV) on days -4 to -2; and undergo TBI on day 0.

TRANSPLANTATION: Patients undergo allogeneic PBSC transplantation on day 0.

GRAFT-VERSUS-HOST-DISEASE (GVHD) PROPHYLAXIS: Patients receive mycophenolate mofetil (MMF) PO every 12 hours on days 0-27 (related donor recipients) or every 8 hours on days 0-96 with taper on day 40 (unrelated donor recipients). Patients also receive cyclosporine IV or PO every 12 hours on days -3 to 56, followed by taper on days 57-180 (related donor recipients) or on days -3 to 100, followed by taper on days 101-177 (unrelated donor recipients).

DONOR LYMPHOCYTE INFUSION: Patients with persistent disease and no GVHD after stopping GVHD prophylaxis receive donor lymphocyte infusion IV over 30 minutes once every 28 days for 3 doses.

Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed up periodically for 2 years and then annually thereafter for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients =< 12 years of age must be approved by Fred Hutchinson Cancer Research Center (FHCRC) principal investigator (PI) in advance
* Patients with a history of Ph+ ALL or CML-BC who, after receiving imatinib mesylate, (or either dasatinib or nilotinib) have < 15% blasts on morphologic marrow evaluation; patients with no detectable Ph+ ALL by morphologic or molecular assays (complete remission) will be accepted
* An appropriately human leukocyte antigen (HLA) matched related or unrelated donor must be prospectively identified who will be available to donate filgrastim (G-CSF) mobilized stem cells
* RELATED DONOR:

  * Related donor who is HLA genotypically identical at least at one haplotype and may be genotypically or phenotypically identical at the allele level at HLA-A, -B, -C, -DRB1, and -DQB1;
  * Donor must consent to G-CSR administration and leukapheresis;
  * Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral, subclavian)
* HLA-MATCHED UNRELATED DONOR:

  * FHCRC matching allowed will be grades 1.0 to 2.1; unrelated donors who are prospectively matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing; only a single allele disparity will be allowed for HLA-A, B, or C as defined by high resolution typing
  * A positive anti-donor cytotoxic crossmatch is an absolute donor exclusion; donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment; this determination is based on the standard practice of the individual institution; the recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain a panel reactive antibody (PRA) screens to class I and class II antigens for all patients before HCT; if the PRA shows >10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained; the donor should be excluded if any of the cytotoxic cross match assays are positive; for those patients with an HLA class I allele mismatch, flow cytometric or B and T cell cytotoxic cross matches should be obtained regardless of the PRA results
  * Patient and donor pairs homozygous at a mismatched allele in the graft rejection vector are considered a two-allele mismatch, i.e., the patient is A*0101 and the donor is A*0102, and this type of mismatch is not allowed
  * Only G-CSF mobilized PBSC only will be permitted as a HSC source on this protocol

Exclusion Criteria:

* Central nervous system (CNS) involvement with leukemia refractory to intrathecal chemotherapy; prior to HSCT (all patients must receive a diagnostic lumbar puncture (LP) with intrathecal (IT) chemotherapy as per standard practice)
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Patients with active non-hematologic malignancies (except non-melanoma skin cancers); this exclusion does not apply to patients with non-hematologic malignancies that do not require therapy
* Patients with a history of non-hematologic malignancies (except non-melanoma skin cancers) currently in a complete remission, who are less than 5 years from the time of complete remission, and have a > 20% risk of disease recurrence; this exclusion does not apply to patients with non-hematologic malignancies that do not require therapy
* Females who are pregnant or breastfeeding
* Patients who are human immunodeficiency virus (HIV)-positive
* Patients with poorly controlled hypertension despite multiple antihypertensives
* Adults: Karnofsky score < 60
* Pediatrics: Lansky play-performance score < 40
* Patients with cardiac ejection fraction < 35% (or, if unable to obtain ejection fraction, shortening fraction of < 26%); ejection fraction is required if age > 50 years or there is a history of anthracycline exposure or history of cardiac disease; patients with a shortening fraction < 26% may be enrolled if approved by a cardiologist
* Diffusing capacity of the lungs for carbon monoxide (DLCO) < 30%
* Total lung capacity (TLC) < 30%
* Forced expiratory volume in one second (FEV1) < 30% and/or receiving supplementary continuous oxygen; the FHCRC PI of the study must approve enrollment of all patients with pulmonary nodules
* Patients with clinical or laboratory evidence of liver disease would be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension; patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, or symptomatic biliary disease
* Creatinine levels more than 2.2 X's the upper limit of normal (ULN) at the laboratory where the analysis was performed
* Patients with active bacterial or fungal infections unresponsive to medical therapy
* For patients receiving dasatinib or nilotinib, baseline corrected QT interval (QTc) (Fridericia's method) prolongation greater than 500 msec
* RELATED DONORS:

  * Identical twin
  * Infection with HIV
  * Inability to achieve adequate venous access
  * Known allergy to G-CSF
  * Current serious system illness
  * Bone marrow (BM) donors
* HLA-MATCHED UNRELATED DONORS:

  * BM donors
  * Donors who are HIV-positive and/or, medical conditions that would result in increased risk for G-CSF mobilization and harvest of PBSC

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2001-07-13 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Georges, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241
- [Derived] Ram R, Storb R, Sandmaier BM, Maloney DG, Woolfrey A, Flowers ME, Maris MB, Laport GG, Chauncey TR, Lange T, Langston AA, Storer B, Georges GE. Non-myeloablative conditioning with allogeneic hematopoietic cell transplantation for the treatment of high-risk acute lymphoblastic leukemia. Haematologica. 2011 Aug;96(8):1113-20. doi: 10.3324/haematol.2011.040261. Epub 2011 Apr 20. PMID 21508120

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Allogeneic Nonmyeloablative HSCT)
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Allogeneic Nonmyeloablative HSCT)
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 57.6 [33.8 to 69.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Relapse Free Survival
Description: Number of patients with relapsed disease within 1 Year post-transplant. Relapse is defined as the detection of > 5% blasts after a documented complete remission.
Time Frame: Assessed up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic Nonmyeloablative HSCT)
Number analyzed (Participants) | 28
Participants | 3

2. Secondary Outcome: Leukemia-free Survival
Description: Number of patients surviving in CR up to five years post-transplant.
Time Frame: Assessed up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic Nonmyeloablative HSCT)
Number analyzed (Participants) | 28
Participants
  6 Months | 19
  1 Year | 17
  2 Years | 13
  3 Years | 11
  4 Years | 11
  5 Years | 10

3. Secondary Outcome: Overall Survival
Description: Number of patients surviving up to five years post-transplant.
Time Frame: Assessed up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic Nonmyeloablative HSCT)
Number analyzed (Participants) | 28
Participants
  6 Months | 26
  1 Year | 24
  2 Years | 19
  3 Years | 17
  4 Years | 16
  5 Years | 13

4. Secondary Outcome: Transplant-related Mortality
Description: Number of patients with TRM within 100 days post-transplant.
Time Frame: At day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic Nonmyeloablative HSCT)
Number analyzed (Participants) | 28
Participants | 1

5. Secondary Outcome: Transplant-related Mortality
Description: Number of patients with TRM within one year post-transplant.
Time Frame: At 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic Nonmyeloablative HSCT)
Number analyzed (Participants) | 28
Participants | 3

ADVERSE EVENTS:
Time Frame: AEs: Conditioning through Day 100; SAEs: Conditioning through Day 200
Arm/Group | Treatment (Allogeneic Nonmyeloablative HSCT)
Serious Adverse Events (participants affected / at risk) | 2/28
Other Adverse Events (participants affected / at risk) | 8/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Allogeneic Nonmyeloablative HSCT) (N=28)
Blood bilirubin increased (Investigations) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Allogeneic Nonmyeloablative HSCT) (N=28)
Anaphylaxis (Immune system disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (3)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes